CLINICAL TRIAL: NCT06202664
Title: Opioid Free Anesthesia for Laparoscopic Cholecystectomy; A Randomized Control Trial at a Tertiary Care Hospital
Brief Title: Opioid Free Anesthesia for Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Muhammad Haroon Anwar (Other Government)
Collaborators: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Muhammad Haroon Anwar, Principal Investigator, Department of Anaesthesia and Critical Care Medicine, Pakistan Institute of Medical Sciences
Organization: Pakistan Institute of Medical Sciences (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F.3-2/2022(ERRB)/PIMS
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Analgesia
Keywords: Opioid Free Anesthesia; Erector Spinae Block; Laparoscopic Cholecystectomy; Intraoperative Hemodynamics; Post operative analgesia
MeSH Terms: conditions — Agnosia | interventions — Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: Patients enrolled will be divided into two groups through computer generated random numbers. Standard ASA monitoring will be done. Intervention will be done at the time of induction of anesthesia that is opioid based analgesia vs Erector Spinae block bilaterally at T6 level. In both groups intra-operative rise in Heart Rate or Blood Pressure or both by more than 20% from baseline value particularly upon skin incision and generation of pneumoperitoneum will indicate inadequate analgesia. This will then be supplemented with 0.5 Mcg/kg of IV Fentanyl increments along with 1g IV Paracetamol and 30 mg IV Ketorolac . Post operatively if VAS score is greater than 4 then rescue analgesia in the form of 1g of IV Paracetamol will be given. This will be supplemented with 15 mg of IV Ketorolac if VAS score is greater than 6. IV Tramadol at dose of 50mg will be given if the VAS score is greater than 8.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid Free Anesthesia Group (Experimental): This will be the experimental group. Patient entering this group through computer generated random numbers will receive opioid free anesthesia in form of ultrasound guided Erector Spinae Block given bilaterally at T6 level.
  Interventions: Procedure: Erector Spinae Block
- Conventional Opioid group (Active Comparator): Patient entering this group through computer generated random numbers will receive opioid based anesthesia.
  Interventions: Drug: Opioid Analgesic

INTERVENTIONS:
Procedure: Erector Spinae Block — Erector Spinae block under ultrasound guidance will be administered bilaterally at T6 level. The block will be administered after induction of general anesthesia with 1mg of IV Midazolam, 2mg/kg of IV Propofol and 0.5 mg/kg of IV Atracurium. After induction patient will be placed in lateral position and then under ultrasound guidance Erector Spinae Block will be administered at T6 level. Drugs administered in the block will include 30ml of 0.25% Bupivacaine and 10ml of 1% Lignocaine (bilaterally). Skin incision for trocar insertion will be given 15 mins after administration of Erector Spinae Block.
  Other Names: Opioid free anesthesia
  Arms: Opioid Free Anesthesia Group
Drug: Opioid Analgesic — This group of patient will receive general anesthesia induction with 1mcg/kg of IV Fentanyl, 2mg/kg of IV Propofol and 0.5 mg/kg of IV Atracurium. 1g of IV paracetamol and 30 mg of IV Ketorolac will be given if intra-operative course suggest inadequate analgesia (Rise in Heart rate ± Blood Pressure by more than 20% from baseline).
  Other Names: Conventional Opioid based analgesia
  Arms: Conventional Opioid group

SUMMARY:
The goal of this interventional study is to check the efficacy of Erector Spinae block as Opioid Free Anesthesia for Laparoscopic Cholecystectomy. Laparoscopic Cholecystectomy is a commonly performed day care procedure. Being a day care procedure the anesthetic technique employed should provide adequate analgesia, allow early mobilization of patient and should mitigate nausea and vomiting which occurs quite frequently in this surgical population. If these goals are achieved patients can be discharged early from hospital setting and this leads to overall cost benefits.

DETAILED DESCRIPTION:
One of the commonest presentations to surgical department is the abdominal pain caused by gall stones. The procedure of choice for treatment of cholelithiasis is Laparoscopic Cholecystectomy; a day care surgical procedure. This is performed under General Anesthesia with Endotracheal tube. During the surgery, anesthetist provides multi-modal analgesia in the form of opioids, NSAIDs and paracetamol. The commonly used Opioids in our setting include Morphine, Fentanyl and Nalbuphine. Opioids provides excellent analgesia but are associated with a number of side effects such as sedation, euphoria or dysphoria, respiratory depression, nausea, vomiting and increase in smooth muscle tone of the gut. These side effects can significantly impair the recovery in post-operative period, leading to prolong hospital stay. As a result opioid free anesthesia could be a suitable alternative to conventional opioid anesthesia for laparoscopic cholecystectomy. By avoiding the adverse effects of opioids; Opioid free anesthesia can lead to early recovery and discharge from the hospital.

One way to provide opioid free anesthesia is by utilizing loco-regional techniques. One of the loco-regional technique which has shown some benefit in laparoscopic cholecystectomy is erector spinae block. However in the available literature the block was utilized for providing post-operative analgesia in laparoscopic cholecystectomy. This Randomized Control Trial will check the efficacy of Erector Spinae Block in providing intra-operative as well as post operative analgesia in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 years to 80 years.
* American Society of Anesthesiologists (ASA) class: I and II.
* Elective Laparoscopic Cholecystectomy under General Anesthesia.
* Duration of surgery being less than 1h

Exclusion Criteria:

* ASA class III or above
* Neuromuscular disease
* Body mass index >35 kg/m2
* known allergy to drugs used in the study
* Ischemic Heart disease, Cardiac Failure, Liver and renal insufficiency
* Intra-operative conversion from laparoscopic to open procedure.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate | Baseline, immediately at/after skin incision, after generation of pneumoperitoneum, and at the end of surgery.
  Heart Rate is measured as a part of standard ASA monitoring through electronic cardiac monitor showing electrocardiogram as well as heart rate (no. of beats/min).
Blood Pressure | Baseline, immediately at/after skin incision, after generation of pneumoperitoneum, and at the end of surgery
  Blood pressure including Systolic, Diastolic and Mean arterial pressure is measured as a part of standard ASA monitoring. This is measured in units of mm of Hg through automated Non-invasive Blood pressure monitoring device.
Post operative pain control | This will be assessed upon patient arrival at Post anesthesia care unit and then 1 hourly interval till 6hours. The pain will be assessed both on rest as well as on cough.
  This will be assessed using Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Intra operative rescue Opioid consumption | Amount of Fentanyl given Intravenously from the time till skin incision to the time at end of surgery
  This will be assessed in terms of micro-grams of Fentanyl consumed intra-operatively in addition to the amount of drug given at induction in control group.
Post operative analgesic consumption | From arrival in the PACU till 6 hours.
  This will be assessed in terms of amount of Tramadol, Ketorolac and Paracetamol consumed in the first 6 hours following surgery as dictated by Visual Analog Scale pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Haroon Anwar, MBBS, Principal Investigator — Department of Anesthesia and Critical Care, Pakistan Institute of Medical Sciences, Islamabad
Locations (1):
- Deparment of Anesthesia and Critical Care Medicine, Pakistan Institute of Medical Sciences, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ragupathy R, Prabhu SCG, Thiyagarajan D, Anto V. Opioid-free anaesthesia for laparoscopic surgeries - A prospective non-randomised study in a tertiary care hospital. Indian J Anaesth. 2022 Mar;66(3):207-212. doi: 10.4103/ija.ija_785_21. Epub 2022 Mar 24. PMID 35497703